CLINICAL TRIAL: NCT03557671
Title: Evaluation of the Hypoallergenicity of a New Formula Based on Hydrolyzed Rice Proteins (TRHF 2017) in Children With Confirmed Immunoglobulin E (IgE) or Non-immunoglobulin E-mediated Cow's Milk Allergy (CMA)
Brief Title: Evaluation of the Hypoallergenicity of a New Formula Based on Hydrolyzed Rice Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Collaborators: Statitec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UP2017-Promyce
Record Dates: First submitted 2018-05-14; First posted 2018-06-15 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRHF - Placebo (Experimental): Each subjects will receive both TRHF and placebo formula during the 1st part of the study
  Interventions: Dietary Supplement: rice formula; Dietary Supplement: placebo
- Placebo - TRHF (Placebo Comparator): Each subjects will receive both TRHF and placebo formula during the 1st part of the study
  Interventions: Dietary Supplement: rice formula; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: rice formula — new rice based thickened formula
Dietary Supplement: placebo — formula previously tolerated by the subject - only for the 1st part of the study

SUMMARY:
The aim of this study is to show the hypoallergenicity of a new thickened rice based formula (TRHF) through a double blind placebo controlled food challenge (DBPCFC), as recommended by the American Academy of Pediatrics, in subjects with IgE-mediated CMA and in subjects with non-IgE-mediated CMA.

DETAILED DESCRIPTION:
The study is made of 2 different steps : 1st step is a double blind randomised food challenge where the new formula is compared to a placebo.

The second part of the trial consists in an open phase during which all infants will be fed with the study formula.

ELIGIBILITY:
Inclusion Criteria:

* with suspected CMA or with a CMA diagnosed by a DBPCFC performed in the last 2 months prior to inclusion
* free of clinical allergic symptoms for at least one week (i.e. successfully fed an elimination diet);
* whose parents signed the informed consent

Exclusion Criteria:

* mainly breast fed, drinking less than 250ml of formula/day, presenting any situation, which, according to the investigator, may interfere with the study participation or lead to a particular risk for the subject

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
hypoallergenicity | 7 days
  the percentage of children tolerating the formula during the double blind placebo controlled food challenge (TRHF 2017 vs. placebo formula).

SECONDARY OUTCOMES:
Regurgitations | 1, 2, 3, 4, 5 and 6 months
  assessed through Vandenplas score ranging from 0 (=less than 2 regurgitation episodes / day) to 6 (=Regurgitation of the complete volume after each feeding)
Vomiting | 1, 2, 3, 4, 5 and 6 months
  (on a 4 level scale)
Abdominal pain | 1, 2, 3, 4, 5 and 6 months
  (severity on a 4 level scale)
Bloating and gas | 1, 2, 3, 4, 5 and 6 months
  (severity on a 4 level scale)
Stool consistency | 1, 2, 3, 4, 5 and 6 months
  assessed through Bristol Stools Form Scale from Type A ( Separate hard lumps, like nuts (hard to pass)) to Type G (Watery, not solid pieces - entirely liquid )
Stool frequency | 1, 2, 3, 4, 5 and 6 months
  (number of stool per day or per week)
Blood in stools | 1, 2, 3, 4, 5 and 6 months
  (presence/absence)
Sleeping time over 24h satisfaction | 1, 2, 3, 4, 5 and 6 months
  (presence/absence)
Unexplained crying | 1, 2, 3, 4, 5 and 6 months
  (yes/no)
Respiratory symptoms | 1, 2, 3, 4, 5 and 6 months
  (severity on a 4 level scale)
Urticaria | 1, 2, 3, 4, 5 and 6 months
  (presence/absence)
Angioedema | 1, 2, 3, 4, 5 and 6 months
  (presence/absence)
Eczema | 1, 2, 3, 4, 5 and 6 months
  severity assessed through SCORAD
Weight | 1, 2, 3, 4, 5 and 6 months
  expressed in kg and in z scores according to the World Health Organization (WHO) Child Growth Standards
Height | 1, 2, 3, 4, 5 and 6 months
  expressed in cm and in z scores according to the WHO Child Growth Standards
BMI | 1, 2, 3, 4, 5 and 6 months
  expressed in value and z scores according to the WHO Child Growth Standards
Head circumference | 1, 2, 3, 4, 5 and 6 months
  expressed in cm and in z scores according to the WHO Child Growth Standards
Number of patients with treatment emergent Adverse Events | 1, 2, 3, 4, 5 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, Study Director — University Federico II
Locations (4):
- CHR Namur, Namur, Belgium
- France (2):
  - Hôpital Saint Vincent de Paul - GHICL, Lille
  - Hopital Trousseau, Paris
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided